CLINICAL TRIAL: NCT04390776
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, CROSS-OVER, SINGLE-DOSE STUDY TO EVALUATE THE BIOEQUIVALENCE OF CANDIDATE CAPSULE FORMULATIONS OF PF-06651600 TO TABLETS AND ESTIMATE THE EFFECT OF HIGH-FAT MEAL ON BIOAVAILABILITY IN HEALTHY PARTICIPANTS
Brief Title: Bioequivalence Study of PF-06651600 Capsules Relative to Tablets and Estimation of Food Effect on Capsules.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981029
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (Experimental): PF-06651600 100 mg Tablets (fasted, Period 1), followed by Capsules (fasted, Period 2), and followed by Capsules (fed, Period 3).
  Interventions: Drug: PF-06651600
- Treatment Sequence 2 (Experimental): PF-06651600 100 mg Capsules (fasted, Period 1), followed by Tablets (fasted, Period 2), and followed by Capsules (fed, Period 3).
  Interventions: Drug: PF-06651600
- Treatment Sequence 3 (Experimental): PF-06651600 100 mg Tablets (fasted, Period 1), followed by Capsules (fasted, Period 2).
  Interventions: Drug: PF-06651600
- Treatment Sequence 4 (Experimental): PF-06651600 100 mg Capsules (fasted, Period 1), followed by Tablets (fasted, Period 2).
  Interventions: Drug: PF-06651600

INTERVENTIONS:
Drug: PF-06651600 — PF-06651600 100 milligrams (mg) will be provided as Tablets and Capsules.

SUMMARY:
The study will be conducted as a Phase 1, open-label, single-dose, randomized, 2- or 3 period, cross over design in a single cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are healthy as determined by medical evaluation including a detailed medical history, complete physical examination, which includes BP and pulse rate measurement, clinical laboratory tests, and cardiac evaluation (including ECG).
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine (including diabetes), pulmonary, gastrointestinal, cardiovascular (including hypertension and congestive heart failure), hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Known immunodeficiency disorder, including positive serology for human immunodeficiency virus (HIV) at screening, or a first degree relative with a hereditary immunodeficiency.

Participants with any of the following acute or chronic infections or infection history:

* Any infection requiring treatment within 2 weeks prior to the dosing visit.
* Any infection requiring hospitalization or parenteral antimicrobial therapy within 60 days of the first dose of study intervention.
* Any infection judged to be an opportunistic infection or clinically significant by the investigator, within the past 6 months of the first dose of study intervention.
* Known active or history of recurrent bacterial, viral, fungal, mycobacterial or other infections.
* History of recurrent (more than one episode of) localized dermatomal herpes zoster, or history of disseminated (single episode) herpes simplex or disseminated herpes zoster.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf)of PF-06651600 | Day 1 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose.
Maximum plasma PF-06651600 concentration (C max) | Day 1 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose.

SECONDARY OUTCOMES:
Single dose time to reach maximum observed plasma concentration (Tmax) of PF-06651600 | Day 1 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose.
Single dose Area under the Curve from Time Zero to Last quantifiable concentration [AUC last) of PF-06651600 | Day 1 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose.
Single dose plasma decay half-life (t 1/2) of PF-06651600 | Day 1 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose.
Single dose Apparent Oral Clearance (CL/F) of PF-06651600 | Day 1 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose.
Single dose Apparent Volume of Distribution (Vz/F) of PF-06651600 | Day 1 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 16 hrs, and Day 2, at 24 hours post-dose.
Frequency of abnormal safety laboratory tests | Baseline up to day 9
Frequency of Adverse Events | Baseline up to day 35

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Saadeddin A, Purohit V, Huh Y, Wong M, Maulny A, Dowty ME, Sagawa K. Virtual Bioequivalence Assessment of Ritlecitinib Capsules with Incorporation of Observed Clinical Variability Using a Physiologically Based Pharmacokinetic Model. AAPS J. 2024 Jan 24;26(1):17. doi: 10.1208/s12248-024-00888-9. PMID 38267790
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981029